CLINICAL TRIAL: NCT04179565
Title: Healthy Children, Healthy Families: Parents Making A Difference: A Randomized Controlled Trial
Brief Title: Healthy Children, Healthy Families: Parents Making A Difference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CornellU
Record Dates: First submitted 2018-09-07; First posted 2019-11-27 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Childhood Obesity Prevention
Keywords: childhood obesity; parenting practices; food and physical activity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Active Comparator): The immediate education (IE) group will receive the intervention, Healthy Children, Healthy Families: Parents Making a Difference! in period 1. In period 2, IE will receive no education and will be followed longitudinally for periods 2 and 3.
  Interventions: Behavioral: Healthy Children Healthy Families
- Delayed intervention (Active Comparator): The delayed education (DE) group will serve as controls in period 1, receiving no intervention. In period 2, the treatments will cross over, so DE will receive the Healthy Children, Healthy Families: Parents Making a Difference! intervention.
  Interventions: Behavioral: Healthy Children Healthy Families

INTERVENTIONS:
Behavioral: Healthy Children Healthy Families — The Healthy Children, Healthy Families: Parents Making a Difference! intervention was developed by the investigators for low-income parents and caregivers focusing on the behaviors most likely to help children avoid unhealthy weight gain.

SUMMARY:
The impacts of Healthy Children, Healthy Families: Parents Making a Difference! (HCHF) on how low-income parents enrolled in the Expanded Food and Nutrition Education Program use effective parenting practices to influence children's healthy eating and active play behavior will be investigated, as compared to a delayed intervention control group.

DETAILED DESCRIPTION:
The Healthy Children, Healthy Families: Parents Making a Difference! (HCHF) curriculum is a Cornell curriculum for parents and caregivers focusing on the behaviors most likely to help children avoid unhealthy weight gain. These behaviors include drinking water or milk instead of sweetened beverages, eating more vegetables and fruits, playing actively, eating fewer high-fat and high-sugar foods, limiting screen time, and having sensible serving sizes. The 8-session curriculum uses a learner-centered dialogue approach, hands-on activities and role plays. The study will include 300 participants with young children 3-5 years old in Head Start and childcare programs in New York City using a randomized control design. In period 1 (9 weeks), half the groups will receive HCHF education (immediate education, IE) and half will serve as controls, receiving no education (delayed education, DE). In period 2 (9 weeks), DE will receive education; IE will receive no education and be followed longitudinally for periods 2 and 3. In period 3 (16 weeks), neither group will receive education and both will be followed longitudinally. Data will be collected at each time point using validated measures, including the HCHF Checklist developed by the investigators and complementary measures that assess parenting feeding practices, food behavior in parents, food behavior in children, and parent self-efficacy around obesity prevention behaviors. It is hypothesized that change pre- to post- HCHF will be greater than control groups, and changes in behavior will be retained post-education.

ELIGIBILITY:
* Inclusion Criteria: Parents/caregivers with young children 3-5 years old
* Exclusion Criteria: Any person who does not have children who are 3-5 years old

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Healthy Children, Healthy Families Checklist | up to 8 months
  The checklist is a 16-item instrument that assesses parents'/caregivers' parenting and personal practices around food and physical activity, as well as the target child's food and physical activity practices. The checklist asks parents to report frequency (per day/week/month) of practices on 5-point Likert-type scales. The constructs measure parent diet quality and physical activity, child diet quality and physical activity, and parenting practices. Each question on the instrument is converted to a numeric value, 1 for the least desirable to 5 for most desirable response. The values for the entire instrument are summed (range 1 - 80 - only those checklists with at least one response are included) and divided by the number of items with a response (0 - 16), resulting in a mean score range of 0 - 5. The questions within each sub-scale are handled in the same way, with a sub-scale range of 0 - 5.
Comprehensive Feeding Practices Questionnaire (CFPQ) | up to 8 months
  Six sub-scales (24 items) aligned with the learning objectives of the intervention, were selected from the original CFPQ. The constructs assessed by the sub-scales include encouraging balance and variety, use of food as reward, parent allowing child to control eating, parental modeling, parental pressure for child to consume more food, and home environment. Response options for 6 items include frequency on a Likert-type scale (never to always) and for 18 items include a Likert scale (strongly disagree to strongly agree). Each response is converted to a numeric value, 1 for the least desirable to 5 for the most desirable option. These values are then summed (range 0 - 120) and divided by the number of items with a response, resulting in a mean scale score range of 0 - 5. The items within each sub-scale are handled in the same way, with the sub-scale ranges of 0 - 5.

SECONDARY OUTCOMES:
Parental self-efficacy | up to 8 months
  Four items were selected assessing parental efficacy for influencing behaviors addressed in the interventions: child's physical activity; and fruit, vegetable, and sugar sweetened beverage intake. The item responses included a 5-point Likert-type scale (not sure to extremely sure). Each question is converted to a numeric value, 1 for the least to 5 for the most desirable. These values are summed (range 0 - 20) and divided by the number of items with a response (0 - 4), resulting in a mean scale score range of 0 - 5.
Food frequency of sugar sweetened beverages and foods | up to 8 months
  Five items were selected from a 10-item instrument; selected items specifically focus on sugar-sweetened beverages and foods with added sugars. Parents report the number of times per day the child consumes each. Based on initial responses, a scoring system was devised that assigned 7 for a response of zero intake (most desirable) to 1 for a response of >2.5 times per day (least desirable). The response values are then summed (range 0 - 35) and divided by 5, resulting in a mean scale score range of 0 - 7.
Parent food choice behaviors | up to 8 months
  Two scales are used from the Food Behavior Checklist to assess parents' self-reported food intake of fruits and vegetables (9 items) and overall diet quality (4 items). Nine items have Likert-type responses with 8 being never to always (scored 1 - 4), and one being poor to excellent (scored 1-5), with the higher score being most desirable in all cases. The responses to two items are no or yes, scored 1 or 5 respectively. Two items ask for number of servings consumed per day and are assigned the value provided. The fruit and vegetable 9-item scale response values are summed (range = 1 - (26+sum of 2 frequency responses). The diet quality 4-item scale response values are summed (range 1 - 17). The sum for each scale is divided by the number of items in the scale resulting in a mean scale score range of 0-7 for the 9-item scale and 0-4.25 for the 4-item scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie S Dollahite, Principal Investigator — Cornell University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2020
Access Criteria: Data access requests will be reviewed by investigators within the Division of Nutritional Sciences at Cornell who were not involved in the study. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Skinner AC, Perrin EM, Skelton JA. Prevalence of obesity and severe obesity in US children, 1999-2014. Obesity (Silver Spring). 2016 May;24(5):1116-23. doi: 10.1002/oby.21497. PMID 27112068
- [Background] Hurley KM, Cross MB, Hughes SO. A systematic review of responsive feeding and child obesity in high-income countries. J Nutr. 2011 Mar;141(3):495-501. doi: 10.3945/jn.110.130047. Epub 2011 Jan 26. PMID 21270360
- [Background] Golley RK, Hendrie GA, Slater A, Corsini N. Interventions that involve parents to improve children's weight-related nutrition intake and activity patterns - what nutrition and activity targets and behaviour change techniques are associated with intervention effectiveness? Obes Rev. 2011 Feb;12(2):114-30. doi: 10.1111/j.1467-789X.2010.00745.x. PMID 20406416
- [Background] Skouteris H, McCabe M, Swinburn B, Newgreen V, Sacher P, Chadwick P. Parental influence and obesity prevention in pre-schoolers: a systematic review of interventions. Obes Rev. 2011 May;12(5):315-28. doi: 10.1111/j.1467-789X.2010.00751.x. PMID 20492538
- [Background] Arnold, C.G. and Sobal, J. 2000. Food practices and nutrition knowledge after graduation from the Expanded Food and Nutrition Education Program (EFNEP). J Nutr Educ Behav. 32:130-138.
- [Background] Auld G, Baker S, Conway L, Dollahite J, Lambea MC, McGirr K. Outcome effectiveness of the widely adopted EFNEP curriculum Eating Smart-Being Active. J Nutr Educ Behav. 2015 Jan-Feb;47(1):19-27. doi: 10.1016/j.jneb.2014.07.001. Epub 2014 Sep 26. PMID 25267324
- [Background] Baral R, Davis GC, Blake S, You W, Serrano E. Using national data to estimate average cost effectiveness of EFNEP outcomes by state/territory. J Nutr Educ Behav. 2013 Mar;45(2):183-7. doi: 10.1016/j.jneb.2012.04.015. Epub 2012 Dec 2. PMID 23211510
- [Background] Brink, M.S. 2000. Expanded food and nutrition education program: A precedent-setting program. Easy Writer Publications.
- [Background] Dollahite J, Kenkel D, Thompson CS. An economic evaluation of the expanded food and nutrition education program. J Nutr Educ Behav. 2008 May-Jun;40(3):134-43. doi: 10.1016/j.jneb.2007.08.011. PMID 18457781
- [Background] Dollahite JS, Pijai EI, Scott-Pierce M, Parker C, Trochim W. A randomized controlled trial of a community-based nutrition education program for low-income parents. J Nutr Educ Behav. 2014 Mar-Apr;46(2):102-9. doi: 10.1016/j.jneb.2013.09.004. Epub 2013 Nov 20. PMID 24268300
- [Background] Agriculture, U.S.D.o., Research, E.a.E., and Scientist, O.o.t.C. 2012. Nutrition and Childhood Obesity Science White Paper.
- [Background] Baranowski T, Cerin E, Baranowski J. Steps in the design, development and formative evaluation of obesity prevention-related behavior change trials. Int J Behav Nutr Phys Act. 2009 Jan 21;6:6. doi: 10.1186/1479-5868-6-6. PMID 19159476
- [Background] Ventura AK, Birch LL. Does parenting affect children's eating and weight status? Int J Behav Nutr Phys Act. 2008 Mar 17;5:15. doi: 10.1186/1479-5868-5-15. PMID 18346282
- [Background] Lent M, Hill TF, Dollahite JS, Wolfe WS, Dickin KL. Healthy children, healthy families: parents making a difference! A curriculum integrating key nutrition, physical activity, and parenting practices to help prevent childhood obesity. J Nutr Educ Behav. 2012 Jan-Feb;44(1):90-2. doi: 10.1016/j.jneb.2011.02.011. Epub 2011 Sep 6. No abstract available. PMID 21900051
- [Background] Dickin KL, Hill TF, Dollahite JS. Practice-based evidence of effectiveness in an integrated nutrition and parenting education intervention for low-income parents. J Acad Nutr Diet. 2014 Jun;114(6):945-950. doi: 10.1016/j.jand.2013.09.029. Epub 2013 Dec 4. PMID 24315130
- [Background] U.S. Department of Agriculture (USDA) & Federal Nutrition Services (FNS). 2016. SNAP-Ed Strategies & Interventions: An obesity Prevention Toolkit for States. Available from:https://snaped.fns.usda.gov/sites/default/files/uploads/NCCORSNAPEdToolkit2016UpdateApril2016FINAL.pdf.
- [Background] Ritchie LD, Welk G, Styne D, Gerstein DE, Crawford PB. Family environment and pediatric overweight: what is a parent to do? J Am Diet Assoc. 2005 May;105(5 Suppl 1):S70-9. doi: 10.1016/j.jada.2005.02.017. PMID 15867900
- [Background] Woodward-Lopez, G., Ritchie, L.D., Gerstein, D.E., and Crawford, P.B. 2006. Obesity: Dietary and developmental influences. Boca Raton: CRC Press.
- [Background] Koplan JP, Liverman CT, Kraak VI; Committee on Prevention of Obesity in Children and Youth. Preventing childhood obesity: health in the balance: executive summary. J Am Diet Assoc. 2005 Jan;105(1):131-8. doi: 10.1016/j.jada.2004.11.023. No abstract available. PMID 15635359
- [Background] Whitaker, R.C.. 2004. A Review of Household Behaviors for Preventing Obesity in Children. Mathematica Policy Research, Inc.: Princeton, NJ.
- [Background] Ontai, L., Ritchie, L.D., Williams, S.T., Young, T., and Townsend, M.S. 2009. Guiding family-based obesity prevention efforts in low-income children in the United States. Part I: What determinants do we target? Int J Child Adolesc health. 2:20-30.
- [Background] Robinson TN. Reducing children's television viewing to prevent obesity: a randomized controlled trial. JAMA. 1999 Oct 27;282(16):1561-7. doi: 10.1001/jama.282.16.1561. PMID 10546696
- [Background] Epstein LH, Valoski AM, Vara LS, McCurley J, Wisniewski L, Kalarchian MA, Klein KR, Shrager LR. Effects of decreasing sedentary behavior and increasing activity on weight change in obese children. Health Psychol. 1995 Mar;14(2):109-15. doi: 10.1037//0278-6133.14.2.109. PMID 7789345
- [Background] Epstein LH, Roemmich JN, Paluch RA, Raynor HA. Influence of changes in sedentary behavior on energy and macronutrient intake in youth. Am J Clin Nutr. 2005 Feb;81(2):361-6. doi: 10.1093/ajcn.81.2.361. PMID 15699222
- [Background] Gortmaker SL, Peterson K, Wiecha J, Sobol AM, Dixit S, Fox MK, Laird N. Reducing obesity via a school-based interdisciplinary intervention among youth: Planet Health. Arch Pediatr Adolesc Med. 1999 Apr;153(4):409-18. doi: 10.1001/archpedi.153.4.409. PMID 10201726
- [Background] Rhee, K. 2008. Childhood overweight and the relationship between parent behaviors, parenting style ' and family functioning. Annals of the American Academy of Political and Social Science. 615:12-37.
- [Background] Clark HR, Goyder E, Bissell P, Blank L, Walters SJ, Peters J. A pilot survey of socio-economic differences in child-feeding behaviours among parents of primary-school children. Public Health Nutr. 2008 Oct;11(10):1030-6. doi: 10.1017/S1368980007001401. Epub 2007 Dec 20. PMID 18093351
- [Background] Institute of Medicine (US) Committee on Prevention of Obesity in Children and Youth; Koplan JP, Liverman CT, Kraak VI, editors. Preventing Childhood Obesity: Health in the Balance. Washington (DC): National Academies Press (US); 2005. Available from http://www.ncbi.nlm.nih.gov/books/NBK83825/ PMID 22379642
- [Background] Davison, K.K. 2004. Activity-related support from parents, peers, and siblings and adolescents' physical activity: are there gender differences? J Phys Act Health. 1:363-376.
- [Background] Horodynski MA, Stommel M. Nutrition education aimed at toddlers: an intervention study. Pediatr Nurs. 2005 Sep-Oct;31(5):364, 367-72. PMID 16295151
- [Background] Beech BM, Klesges RC, Kumanyika SK, Murray DM, Klesges L, McClanahan B, Slawson D, Nunnally C, Rochon J, McLain-Allen B, Pree-Cary J. Child- and parent-targeted interventions: the Memphis GEMS pilot study. Ethn Dis. 2003 Winter;13(1 Suppl 1):S40-53. PMID 12713210
- [Background] Haire-Joshu D, Elliott MB, Caito NM, Hessler K, Nanney MS, Hale N, Boehmer TK, Kreuter M, Brownson RC. High 5 for Kids: the impact of a home visiting program on fruit and vegetable intake of parents and their preschool children. Prev Med. 2008 Jul;47(1):77-82. doi: 10.1016/j.ypmed.2008.03.016. Epub 2008 Apr 9. PMID 18486203
- [Background] Harvey-Berino J, Rourke J. Obesity prevention in preschool native-american children: a pilot study using home visiting. Obes Res. 2003 May;11(5):606-11. doi: 10.1038/oby.2003.87. PMID 12740449
- [Background] Cullen KW, Lara Smalling A, Thompson D, Watson KB, Reed D, Konzelmann K. Creating healthful home food environments: results of a study with participants in the expanded food and nutrition education program. J Nutr Educ Behav. 2009 Nov-Dec;41(6):380-8. doi: 10.1016/j.jneb.2008.12.007. PMID 19879493
- [Background] New York State Department of Health. 2016. Eat Well Play hard in Child Care Settings. Available from: http://www.health.ny.gov/prevention/nutrition/cacfp/ewphccs.
- [Background] Gabor V, Cates S, Gleason S, Long V, Aponte Clarke G, Blitstein J. 2012. SNAP education and evaluation (wave I): final report. Available from: http://www.fns.usda.gov/ snap-education-and-evaluation-study-wave-i.
- [Background] Food Trust. 2007. Kindergarten Initiative: A Healthy Start to a Healthy Life, 2007: Philadelphia PA: A Report of the Food Trust.
- [Background] Food Trust. 2010. Intervention: The Kindergarten Initiative. Available from: http://centertrt.org/content/docs/intervention_documents/intervention_templates/kindergarten_intitiative_template.pdf.
- [Background] National Heart, Lung, and Blood Institute. 2016. We Can! Ways to Enhance Children's Activity & Nutrition. Available from: http://www.nhlbi.nih.gov/health/educational/wecan/
- [Background] Grutzmacher, S. 2013. Text2BHealthy: A case study of planning, implementing, and evaluating a targeted text-based nutrition education program 141st APHA Annual Meeting and Exposition. APHA.
- [Background] Speirs KE, Grutzmacher SK, Munger AL, Messina LA. Recruitment and retention in an SMS-based health education program: Lessons learned from Text2BHealthy. Health Informatics J. 2016 Sep;22(3):651-8. doi: 10.1177/1460458215577995. Epub 2015 Apr 27. PMID 25916832
- [Background] Arnold, C.G. and Sobal, J. 2000. Food practices and nutrition knowledge after graduation from the Expanded Food and Nutrition Education Program (EFNEP). J Nutr Educ. 32:130-138.
- [Background] Amstutz, M.K., Dixon, D.L. 1986. Dietary changes resulting from the Expanded Food and Nutrition Education Program. J Nutr Educ. 18:55-60.
- [Background] Nierman, L.G., A longitudinal study of the retention of foods and nutrition knowledge and practices of participants from the Michigan Expanded Food and Nutrition Education Program, 1986, Michigan State University: East Lansing, MI.
- [Background] Wardlaw, M. and Baker, S. 2012. Long-term evaluation of EFNEP and SNAP-Ed. Forum Fam Consum Issues.17 (2) Retrieved from http://ncsu. edu/ffci/publications/2012/v17-n2-2012-summer-fall/wardl.
- [Background] Norris, J. 2003. From Telling to Teaching: A Dialogue Approach to Adult Learning. Featuring a Step-by-step Workshop Design Model that Will Transform You, Your Teaching, and Your Learners! North Myrtle Beach, NC: Learning By Dialogue.
- [Background] Bandura, A. 1986. Social Foundations of Thought and Action: A Social Cognitive Theory. Prentice-Hall, Inc.
- [Background] Ryan, R.M., Patrick, H., Deci, E.L., and Williams, G.C. 2008. Facilitating health behaviour change and its maintenance: Interventions based on self-determination theory. European Health Psychologist. 10:2-5.
- [Background] Oliveria SA, Ellison RC, Moore LL, Gillman MW, Garrahie EJ, Singer MR. Parent-child relationships in nutrient intake: the Framingham Children's Study. Am J Clin Nutr. 1992 Sep;56(3):593-8. doi: 10.1093/ajcn/56.3.593. PMID 1503074
- [Background] van der Horst K, Oenema A, Ferreira I, Wendel-Vos W, Giskes K, van Lenthe F, Brug J. A systematic review of environmental correlates of obesity-related dietary behaviors in youth. Health Educ Res. 2007 Apr;22(2):203-26. doi: 10.1093/her/cyl069. Epub 2006 Jul 21. PMID 16861362
- [Background] Cullen KW, Baranowski T, Rittenberry L, Cosart C, Hebert D, de Moor C. Child-reported family and peer influences on fruit, juice and vegetable consumption: reliability and validity of measures. Health Educ Res. 2001 Apr;16(2):187-200. doi: 10.1093/her/16.2.187. PMID 11345661
- [Background] Fisher JO, Mitchell DC, Smiciklas-Wright H, Birch LL. Parental influences on young girls' fruit and vegetable, micronutrient, and fat intakes. J Am Diet Assoc. 2002 Jan;102(1):58-64. doi: 10.1016/s0002-8223(02)90017-9. PMID 11794503
- [Background] Wardle J, Carnell S, Cooke L. Parental control over feeding and children's fruit and vegetable intake: how are they related? J Am Diet Assoc. 2005 Feb;105(2):227-32. doi: 10.1016/j.jada.2004.11.006. PMID 15668680
- [Background] Raudsepp, L. and Viira, R. 2000. Influence of parents' and siblings' physical activity on activity levels of adolescents. Eur J Phys Educ. 5:169-178.
- [Background] Trost SG, Kerr LM, Ward DS, Pate RR. Physical activity and determinants of physical activity in obese and non-obese children. Int J Obes Relat Metab Disord. 2001 Jun;25(6):822-9. doi: 10.1038/sj.ijo.0801621. PMID 11439296
- [Background] Reimer K, Smith C, Reicks M, Henry H, Thomas R, Atwell J. Child-feeding strategies of African American women according to stage of change for fruit and vegetable consumption. Public Health Nutr. 2004 Jun;7(4):505-12. doi: 10.1079/PHN2003551. PMID 15153256
- [Background] Chapman-Novakofski K, Karduck J. Improvement in knowledge, social cognitive theory variables, and movement through stages of change after a community-based diabetes education program. J Am Diet Assoc. 2005 Oct;105(10):1613-6. doi: 10.1016/j.jada.2005.07.010. PMID 16183364
- [Background] Schnoll R, Zimmerman BJ. Self-regulation training enhances dietary self-efficacy and dietary fiber consumption. J Am Diet Assoc. 2001 Sep;101(9):1006-11. doi: 10.1016/S0002-8223(01)00249-8. PMID 11573751
- [Background] Shannon J, Kirkley B, Ammerman A, Keyserling T, Kelsey K, DeVellis R, Simpson RJ Jr. Self-efficacy as a predictor of dietary change in a low-socioeconomic-status southern adult population. Health Educ Behav. 1997 Jun;24(3):357-68. doi: 10.1177/109019819702400308. PMID 9158979
- [Background] Townsend MS, Kaiser LL. Development of a tool to assess psychosocial indicators of fruit and vegetable intake for 2 federal programs. J Nutr Educ Behav. 2005 Jul-Aug;37(4):170-84. doi: 10.1016/s1499-4046(06)60243-1. PMID 16029687
- [Background] Kristal AR, Glanz K, Tilley BC, Li S. Mediating factors in dietary change: understanding the impact of a worksite nutrition intervention. Health Educ Behav. 2000 Feb;27(1):112-25. doi: 10.1177/109019810002700110. PMID 10709796
- [Background] Henry H, Reimer K, Smith C, Reicks M. Associations of decisional balance, processes of change, and self-efficacy with stages of change for increased fruit and vegetable intake among low-income, African-American mothers. J Am Diet Assoc. 2006 Jun;106(6):841-9. doi: 10.1016/j.jada.2006.03.012. PMID 16720125
- [Background] Delahanty LM, Conroy MB, Nathan DM; Diabetes Prevention Program Research Group. Psychological predictors of physical activity in the diabetes prevention program. J Am Diet Assoc. 2006 May;106(5):698-705. doi: 10.1016/j.jada.2006.02.011. PMID 16647327
- [Background] Fahrenwald NL, Walker SN. Application of the Transtheoretical Model of behavior change to the physical activity behavior of WIC mothers. Public Health Nurs. 2003 Jul-Aug;20(4):307-17. doi: 10.1046/j.1525-1446.2003.20408.x. PMID 12823791
- [Background] Dix T. The affective organization of parenting: adaptive and maladaptive processes. Psychol Bull. 1991 Jul;110(1):3-25. doi: 10.1037/0033-2909.110.1.3. PMID 1891517
- [Background] Satter, E. 2005. Your Child's Weight: Helping Without Harming. Madison, WI: Kelcy Press.
- [Background] Hughes SO, Power TG, Orlet Fisher J, Mueller S, Nicklas TA. Revisiting a neglected construct: parenting styles in a child-feeding context. Appetite. 2005 Feb;44(1):83-92. doi: 10.1016/j.appet.2004.08.007. Epub 2004 Nov 13. PMID 15604035
- [Background] Sallis JF, Alcaraz JE, McKenzie TL, Hovell MF, Kolody B, Nader PR. Parental behavior in relation to physical activity and fitness in 9-year-old children. Am J Dis Child. 1992 Nov;146(11):1383-8. doi: 10.1001/archpedi.1992.02160230141035. PMID 1415081
- [Background] Davison KK, Cutting TM, Birch LL. Parents' activity-related parenting practices predict girls' physical activity. Med Sci Sports Exerc. 2003 Sep;35(9):1589-95. doi: 10.1249/01.MSS.0000084524.19408.0C. PMID 12972881
- [Background] Bungum TJ, Vincent ML. Determinants of physical activity among female adolescents. Am J Prev Med. 1997 Mar-Apr;13(2):115-22. PMID 9088448
- [Background] Brustad. 1993. Who will go out and play? Parental and psychological influences on children's attraction to physical activity. Pediatr Exerc Sci. 5:210-223.
- [Background] Golan M, Weizman A. Reliability and validity of the Family Eating and Activity Habits Questionnaire. Eur J Clin Nutr. 1998 Oct;52(10):771-7. doi: 10.1038/sj.ejcn.1600647. PMID 9805227
- [Background] Cullen KW, Baranowski T, Owens E, Marsh T, Rittenberry L, de Moor C. Availability, accessibility, and preferences for fruit, 100% fruit juice, and vegetables influence children's dietary behavior. Health Educ Behav. 2003 Oct;30(5):615-26. doi: 10.1177/1090198103257254. PMID 14582601
- [Background] Nicklas TA, Baranowski T, Baranowski JC, Cullen K, Rittenberry L, Olvera N. Family and child-care provider influences on preschool children's fruit, juice, and vegetable consumption. Nutr Rev. 2001 Jul;59(7):224-35. doi: 10.1111/j.1753-4887.2001.tb07014.x. PMID 11475448
- [Background] Hearn, M., T., B., J., B., Doyle, C., Smith, M., Lin, L.S., and Resnicow, K. 1998. Environmental influences on dietary behavior among children: availability and accessibility of fruit and vegetables enable consumption. J Health Educ. 29:26-32.
- [Background] Cullen KW, Eagan J, Baranowski T, Owens E, de Moor C. Effect of a la carte and snack bar foods at school on children's lunchtime intake of fruits and vegetables. J Am Diet Assoc. 2000 Dec;100(12):1482-6. doi: 10.1016/s0002-8223(00)00414-4. PMID 11138440
- [Background] Brown KA, Ogden J, Vogele C, Gibson EL. The role of parental control practices in explaining children's diet and BMI. Appetite. 2008 Mar-May;50(2-3):252-9. doi: 10.1016/j.appet.2007.07.010. Epub 2007 Aug 1. PMID 17804116
- [Background] Ogden J, Reynolds R, Smith A. Expanding the concept of parental control: a role for overt and covert control in children's snacking behaviour? Appetite. 2006 Jul;47(1):100-6. doi: 10.1016/j.appet.2006.03.330. Epub 2006 May 8. PMID 16682098
- [Background] Spurrier NJ, Magarey AA, Golley R, Curnow F, Sawyer MG. Relationships between the home environment and physical activity and dietary patterns of preschool children: a cross-sectional study. Int J Behav Nutr Phys Act. 2008 May 30;5:31. doi: 10.1186/1479-5868-5-31. PMID 18513416
- [Background] Dickin KL, Larios F, Parra PA. Cognitive Interviewing to Enhance Comprehension and Accuracy of Responses to a Spanish-Language Nutrition Program Evaluation Tool. J Nutr Educ Behav. 2015 Sep-Oct;47(5):465-71.e1. doi: 10.1016/j.jneb.2015.06.008. Epub 2015 Jul 22. PMID 26209887
- [Background] Dickin KL, Lent M, Lu AH, Sequeira J, Dollahite JS. Developing a measure of behavior change in a program to help low-income parents prevent unhealthful weight gain in children. J Nutr Educ Behav. 2012 Jan-Feb;44(1):12-21. doi: 10.1016/j.jneb.2011.02.015. Epub 2011 Oct 13. PMID 21996430
- [Background] U.S. Department of Agriculture (USDA), Nutrition Evaluation Reporting System (NEERS5), 2009, Cooperative State Research, Education, and Extension Service, USDA.
- [Background] Musher-Eizenman D, Holub S. Comprehensive Feeding Practices Questionnaire: validation of a new measure of parental feeding practices. J Pediatr Psychol. 2007 Sep;32(8):960-72. doi: 10.1093/jpepsy/jsm037. Epub 2007 May 28. PMID 17535817
- [Background] Wright JA, Adams WG, Laforge RG, Berry D, Friedman RH. Assessing parental self-efficacy for obesity prevention related behaviors. Int J Behav Nutr Phys Act. 2014 Apr 22;11:53. doi: 10.1186/1479-5868-11-53. PMID 24750693
- [Background] Murphy SP, Kaiser LL, Townsend MS, Allen LH. Evaluation of validity of items for a food behavior checklist. J Am Diet Assoc. 2001 Jul;101(7):751-61. doi: 10.1016/S0002-8223(01)00189-4. PMID 11478471
- [Background] Koleilat M, Whaley SE. Reliability and Validity of Food Frequency Questions to Assess Beverage and Food Group Intakes among Low-Income 2- to 4-Year-Old Children. J Acad Nutr Diet. 2016 Jun;116(6):931-9. doi: 10.1016/j.jand.2016.02.014. Epub 2016 Mar 31. PMID 27050726
- [Background] Dickin KL, Seim G. Adapting the Trials of Improved Practices (TIPs) approach to explore the acceptability and feasibility of nutrition and parenting recommendations: what works for low-income families? Matern Child Nutr. 2015 Oct;11(4):897-914. doi: 10.1111/mcn.12078. Epub 2013 Sep 13. PMID 24028083